CLINICAL TRIAL: NCT07031284
Title: Cardiac Magnetic Resonance in Patients With Giant Cell Arteritis
Brief Title: Cardiac Involvement in Patients With Giant Cell Arteritis
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Isaak, Radiologist, , Radiology Clinic, University Hospital, Bonn
Other Study IDs: 2020-475-BON
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Cardiac Magnetic Resonance Imaging; Giant Cell Arteritis; Cardiovascular Disease; Tissue Characterization; Myocardial Disease
MeSH Terms: conditions — Giant Cell Arteritis; Cardiovascular Diseases; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with diagnosed GCA: Clinically diagnosed GCA-patients from the Department of Rheumatology.
- Healthy controls: Healthy control group from historical data

SUMMARY:
This prospective observational study aims to investigate whether patients with newly diagnosed giant cell arteritis (GCA) show signs of cardiac involvement. Using multiparametric cardiac magnetic resonance imaging (CMR), functional, structural, and tissue-specific cardiac parameters are assesed. All participants undergo CMR at baseline and a follow up CMR after approximately six months. Healthy controls are included for comparison. Results may help improve early detection and monitoring of cardiovascular complications in GCA.

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) is a systemic inflammatory vasculitis of older adults, potentially involving the cardiovascular system. While aortic and vascular complications are well described, myocardial involvement remains understudied and often subclinical. GCA is associated with increased all-cause mortality and cardiovascular disease, therefore early detection of cardiovascular involvement is essential.

This prospective single-center study investigates myocardial tissue alterations in patients with newly diagnosed GCA using comprehensive multiparametric cardiac magnetic resonance imaging (CMR). All participants gave written informed consent prior to cardiac MRI. Diagnosis of GCA was established according to current clinical and ultrasound criteria. Only subjects without general contraindications for contrast-enhanced CMR were included (e.g., MRI-incompatible implants, known allergy to MRI contrast agents, severe renal impairment, brestfeeding, pregnancy, and claustrophobia). The CMR protocol includes native T1- and post contrast T1-, T2 mapping, late gadolinium enhancement (LGE), T2-weighted short-tau inversion-recovery sequences and functional cine imaging.

The study comprises a baseline CMR and a follow-up scan after approximately 6 months. The extracellular volume fraction (ECV) is calculated from pre and post-contrast T1-mapping and current hematocrit. Left and right ventricular function and volumes were assessed on short-axis cine images. Functional parameters were indexed to body surface area. Imaging results are correlated with inflammatory markers and clinical features. A healthy control group from historiacal datasets is used for comparison. Group comparisons are performed using t-tests, Mann-Whitney U, and chi-square tests; paired t-tests assessed longitudinal changes.

The study aims to evaluate the prevalence, pattern, and evolution of cardiac changes in GCA and explore their clinical relevance for cardiovascular risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed GCA

Exclusion Criteria:

* MRI contraindications (e.g. non-compartible pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 GCA-diagnosed patients (mean age 73 years, SD 9; 42% female)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Differences in myocardial mapping between GCA patients and a healthy control | Baseline Cardiac MRI was performed in an avarage of 31 days after first symptoms
  Quantitative assessment of native myocardial T1, T2, and extracellular volume (ECV) by cardiac MRI at baseline to evaluate subclinical myocardial involvement in patients with newly diagnosed giant cell arteritis compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Petzinna, Dr., Principal Investigator — University Hospital Bonn, Department of Rheumatology; Alexander Isaak, PD Dr., Principal Investigator — University Hospital Bonn, Department of Radiology; Julian Luetkens, Prof. Dr., Study Director — University Hospital Bonn, Department of Radiology
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided